CLINICAL TRIAL: NCT00185679
Title: A Feasibility Study Evaluating Haploidentical Allogeneic Transplantation Using the CliniMACS System in Patients With Advanced Hematologic Malignancies
Brief Title: Haploid Allogeneic Transplant Using the CliniMACS System
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This study was superseded by the subsequent study IRB-15919 (NCT01050764)
Sponsor: Ginna Laport (Other)
Responsible Party: Sponsor-Investigator, Ginna Laport, Associate Professor of Medicine, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-12600; BMT123 (Other: OnCore); NCI-2011-00424 (Other: NCI PDQ); 77453 (Other: Historic IRB SQL database number)
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Results first posted 2015-03-09 (Estimated); Last update posted 2015-03-09 (Estimated); Status verified 2015-02

CONDITIONS: Acute Myelogenous Leukemia (AML) - Relapsed, Primary Refractory Disease or Poor Risk Factors; Chronic Myelogenous Leukemia (CML) - Accelerated or Second Chronic Phase; Myelodysplastic Syndrome (MDS) - High and Intermediate Risk; Non-Hodgkin's Lymphoma (NHL); Chronic Lymphocytic Leukemia (CLL) - Refractory
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Recurrence; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Myelodysplastic Syndromes; Lymphoma, Non-Hodgkin; Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Haploidentical Allogeneic Transplant Using CliniMACS System (Experimental): The CliniMACS cell selection system (Miltenyi Biotec) will be used to enrich hematopoietic stem cells from related, haploidentical, HLA-matched donors, who matched on the A,B,C and DRB1, DQ loci.
  Interventions: Device: CliniMACS System

INTERVENTIONS:
Device: CliniMACS System — The CliniMACS System is a cell selection device consisting of the following components:
  1. Computer-controlled instrument;
  2. Sterile disposable tubing set (PVC tubing, filters and bags connected to two separation columns containing an iron/plastic matrix)
  3. Anti-CD34 antibody reagent (murine monoclonal antibody chemically coupled to a magnetic particle)
  4. Wash buffer
  Other Names: CliniMACS Cell Selection System

SUMMARY:
To assess the proportion of patients with donor neutrophil engraftment within 30 days of allogeneic transplant. To assess the incidence of acute GvHD during the first 100 days after transplantation.

DETAILED DESCRIPTION:
To assess the proportion of patients with donor neutrophil engraftment within 30 days of allogeneic transplant; assess the incidence of acute GvHD during the first 100 days after transplantation; and assess platelet engraftment, graft failure, chronic GvHD, clinical safety, and devise performance.

ELIGIBILITY:
RECIPIENT INCLUSION CRITERIA

Histopathologically-confirmed diagnosis of hematological or lymphatic malignancy, defined as one of the following:

* Acute myeloid leukemia (AML) as primary refractory disease, or in relapse
* Acute leukemia in first remission with poor risk factors and molecular prognosis
* AML with -5,-7, t(6;9), tri8, -11
* Acute lymphocytic / lymphoblastic leukemia (ALL) with Phil+ t(9;22),(q34;q11.2), and t(4:11)(q21;23)
* Chronic myelogenous leukemia (CML in accelerated, second chronic phase
* Myelodysplastic syndrome with high intermediate to high risk categories
* Non-Hodgkin's lymphoma (NHL)
* Chronic lymphocytic leukemia (CLL), Refractory < 50 years old at time of registration Donor is related Donor is genotypically-matched and haploidentical for HLA-A, B,C and DRB1, DQ loci Donor differs for 2 or 3 HLA alleles on the unshared haplotype in the GvHD direction No HLA-matched sibling or matched unrelated donor is identified ECOG performance status not more than 2 LVEF > 45% DLCO > 50% corrected for hemoglobin Serum creatinine
* < 1.5 mg/dL OR
* creatinine clearance > 50 mL/min for those above serum creatinine of 1.5 mg/dL serum bilirubin < 2.0 mg/dL ALT < 2x ULN (unless secondary to disease) Females of childbearing potential must have a negative serum or urine beta-HCG test within 3 weeks of registration No prior cancer within 5 years with the exception of surgically-cured, non-melanoma skin cancer or in situ cancer of the cervix No prior myeloablative therapy or transplant Duly-executed informed consent

RECIPIENT EXCLUSION CRITERIA Suitable candidate for autologous transplantation Participation in other investigational drugs or devices trials that might influence the study endpoints Evidence of active hepatitis Evidence of active cirrhosis HIV-positive History of invasive aspergillosis Presence of any other uncontrolled, active infection, ie, bacterial, viral or fungal Uncontrolled CNS involvement Documented allergy to murine proteins Documented allergy to iron dextran Lactating female Female of child-bearing potential unwilling to implement adequate birth control Medical problem / neurologic/psychiatric dysfunction which would impair his/her ability to be compliant with the medical regimen and/or to tolerate transplantation, in the opinion of the principal investigator Medical problem / neurologic/psychiatric dysfunction which would prolong hematologic recovery and place the recipient at unacceptable risk, in the opinion of the principal investigator would .

DONOR INCLUSION CRITERIA Age < 60 years Weight > 25 kg Medical history and physical examination confirm good health status as defined by institutional standards Within 30 days of apheresis collection, seronegative for HIV assessed as HIV Ag; HIV 1+2 Ab; or HTLV I/II Ab Within 30 days of apheresis collection, seronegative for hepatitis assessed as HBsAg; HBcAb (IgM and IgG); or HCV Ab Within 30 days of apheresis collection, seronegative for syphilis assessed as RPR Genotypically haploidentical as determined by HLA typing Female donors of child-bearing potential must have a negative serum or urine beta-HCG test within 3 weeks of mobilization Capable of undergoing leukapheresis Has adequate venous access Willing to undergo insertion of a central catheter should leukapheresis via peripheral vein be inadequate Agreeable to second donation of PBPC (or a bone marrow harvest) should the recipient fail to demonstrate sustained engraftment following the transplant Duly-executed informed consent Screened for CMV seroreactivity

* Must be seronegative donor if recipeint is seronegative.
* Otherwise the donor will be selected on the ability of NK cell alloreactivity based upon HLA typing results and donors who are capable of NK cell alloreactivity will be used preferentially.

DONOR EXCLUSION CRITERIA Evidence of active infection (including urinary tract infection, or upper respiratory tract infection) Evidence of hepatitis (on screening) Medical, physical or psychological reason which makes the donor unlikely to tolerate or cooperate with growth factor therapy and leukapheresis Factors placing donor at increased risk for leukapheresis or G-CSF-related complications Lactating female Female of child-bearing potential unwilling to implement adequate birth control HIV-positive

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2001-11; Primary Completion 2009-10 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ginna G Laport, MD, Principal Investigator — Stanford Cancer Institute
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Haploidentical Allogeneic Transplant Using CliniMACS System: The CliniMACS cell selection system (Miltenyi Biotec) will be used to enrich hematopoietic stem cells from related, haploidentical, HLA-matched donors, who matched on the A,B,C and DRB1, DQ loci.
  CliniMACS System: The CliniMACS System is a cell selection device consisting of the following components:
  1. Computer-controlled instrument;
  2. Sterile disposable tubing set (PVC tubing, filters and bags connected to two separation columns containing an iron/plastic matrix)
  3. Anti-CD34 antibody reagent (murine monoclonal antibody chemically coupled to a magnetic particle)
  4. Wash buffer
Period: Overall Study
Arm/Group | Haploidentical Allogeneic Transplant Using CliniMACS System
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Haploidentical Allogeneic Transplant Using CliniMACS System: The CliniMACS cell selection system (Miltenyi Biotec) will be used to enrich hematopoietic stem cells from related, haploidentical, HLA-matched donors, who matched on the A,B,C and DRB1, DQ loci.
  The CliniMACS System is a cell selection device consisting of the following components:
  1. Computer-controlled instrument;
  2. Sterile disposable tubing set (PVC tubing, filters and bags connected to two separation columns containing an iron/plastic matrix)
  3. Anti-CD34 antibody reagent (murine monoclonal antibody chemically coupled to a magnetic particle)
  4. Wash buffer
Arm/Group | Haploidentical Allogeneic Transplant Using CliniMACS System
Number analyzed (Participants) | 13
Age, Continuous [Median (Full Range); unit: years] | 27 [21 to 51]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 7

OUTCOME MEASURES:

1. Primary Outcome: Neutrophil Engraftment
Description: Number of subjects recovering neutrophils, assessed as 1st of 3 consecutive days on which ANC > 0.5x10e9/L
Time Frame: 30 days post-transplant
Measure: Number; unit: participants
Arm/Group | Haploidentical Allogeneic Transplant Using CliniMACS System
Number analyzed (Participants) | 13
participants | 12

2. Secondary Outcome: Acute GvHD (Grade II-IV)
Description: Number of subjects with acute GvHD (grade II-IV) within 100 days post-transplant, per the Consensus Conference on Acute GvHD Grading (Przepiorka D, et al. Bone Marrow Transplantation. 1995. 15:825-828).
Time Frame: within 100 days post-transplant
Measure: Number; unit: participants
Arm/Group | Haploidentical Allogeneic Transplant Using CliniMACS System
Number analyzed (Participants) | 13
participants | 1

3. Secondary Outcome: Platelet Recovery
Description: Number of subjects recovering platelets to > 20x10e9/L, assessed on the 7th day unsupported by platelet transfusions
Time Frame: 40 days
Measure: Number; unit: participants
Arm/Group | Haploidentical Allogeneic Transplant Using CliniMACS System
Number analyzed (Participants) | 13
participants | 12

ADVERSE EVENTS:
Time Frame: SAEs reported through Day 100 post-transplant.
Description: Non-serious adverse events not reported
Arm/Group | Haploidentical Allogeneic Transplant Using CliniMACS System
Serious Adverse Events (participants affected / at risk) | 3/13
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Haploidentical Allogeneic Transplant Using CliniMACS System (N=13)
Treatment-related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Infections and infestations - Other, demyelinating ecephalitis (Infections and infestations) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, pulmonary fungal infection (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Death NOS - Other, graft failure (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No